CLINICAL TRIAL: NCT00576771
Title: Effects of Different Assisted Mechanical Ventilation in ALI/ARDS Patients: PSV, NAVA and Controlled by Patient
Brief Title: Effects of Different Assisted Mechanical Ventilation in Acute Lung Injury/Acute Respiratory Distress Syndrome (ALI/ARDS) Patients: Pressure Support Ventilation (PSV), Neurally Adjusted Ventilatory Assist (NAVA) and Controlled by Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 222222
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: ALI/ARDS Patients
MeSH Terms: interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): ALI/ARDS patients
  evaluated the effect of PSV, NAVA and assisted controlled mechanical ventilation by patient through a button
  Interventions: Procedure: PSV; Procedure: NAVA; Procedure: patient-controlled

INTERVENTIONS:
Procedure: PSV — Pressure Support Ventilation
Procedure: NAVA — Neurally Adjusted Ventilatory Assist
Procedure: patient-controlled — assisted controlled MV through a button

SUMMARY:
The investigators' aim is to study the effect of pressure support ventilation versus neurally adjusted assist (NAVA) and controlled by patient in mechanically ventilated ALI/ARDS subjects.

DETAILED DESCRIPTION:
In this study, PSV is compared with NAVA and assisted mechanically ventilation controlled by patient through a button. Inclusion criteria are: assisted mechanically ventilated ALI/ARDS patients.

ELIGIBILITY:
Inclusion Criteria:

* ALI/ARDS patients

Exclusion Criteria:

* Haemodynamic instability
* Barotrauma
* COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Respiratory mechanics work of breathing,end expiratory lung volume, gas exchange, dead space, patient's comfort level | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Policlinico Hospital
Locations (1):
- Policlinico Hospital, Milan, Italy